CLINICAL TRIAL: NCT06164379
Title: A Double-blind, Randomized Controlled Study of Finerenone vs. Spironolactone in Hypertensive Patients With Primary Aldosteronism
Brief Title: Efficacy and Safety of Finerenone vs. Spironolactone in Patients With Primary Aldosteronism
Acronym: FAVOR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji-Guang Wang, Director of the Shanghai Institute of Hypertension, Director of the Department of Hypertension, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FAVOR
Record Dates: First submitted 2023-12-02; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Primary Aldosteronism
Keywords: Primary Aldosteronism; Spironolactone; Finerenone
MeSH Terms: conditions — Hyperaldosteronism | interventions — finerenone; Spironolactone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Finerenone group (Experimental): After the induction period of two weeks, the patients with primary aldosteronism were randomized in an equal ratio to receive finerenone 10mg once daily. Patients received the initial dose (10mg, week 0) of drug for the first two weeks of randomized treatments period. Thereafter, the dose of finerenone would not be changed for the adequate blood pressure (BP) control and the normal serum potassium. For patients not meeting BP < 140/90mmHg and the serum potassium ≥ 3.5 mmol/L, the dose of finerenone would be increased to 20mg once daily for the second 2 weeks later (week 2) and 30 mg 4 weeks later (week 4), respectively. The whole treatment period was 8 weeks. if blood pressure > 160/110 mmHg during the clinical trial, amlodipine 5 mg once was added.
  Interventions: Drug: Finerenone
- Spironolactone group (Active Comparator): After the induction period of two weeks, the patients with primary aldosteronism were randomized in an equal ratio to receive spironolactone 20mg once daily. Patients received the initial dose (20mg, week 0) of drug for the first two weeks of randomized treatments period. Thereafter, the dose of spironolactone would not be changed for the adequate blood pressure (BP) control and the normal serum potassium. For patients not meeting BP < 140/90mmHg and the serum potassium ≥ 3.5 mmol/L, the dose of finernone would be increased to 40mg once daily for the second 2 weeks later (week 2) and 60 mg 4 weeks later (week 4), respectively. the whole treatment period was 8 weeks. if blood pressure > 160/110 mmHg during the clinical trial, amlodipine 5 mg once was added.
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Finerenone — At every visit, the clinic and ambulatory blood pressure will be measured. The levels of serum potassium, creatinine, renin, aldosterone will be examined. The urinary microalbumin creatinine ratio will be also examined.
  Arms: Finerenone group
Drug: Spironolactone — At every visit, the clinic and ambulatory blood pressure will be measured. The levels of serum potassium, creatinine, renin, aldosterone will be examined. The urinary microalbumin creatinine ratio will be also examined.
  Arms: Spironolactone group

SUMMARY:
To study the efficacy and safety of finerenone vs. spironolactone in patients with primary aldosteronism

DETAILED DESCRIPTION:
1. Study design: This is a multi-center, double-blind, randomized, non-inferiority trial of finerenone vs. spironolactone in hypertensive patients with primary aldosteronism (PA). All patients will be randomized into finerenone group (Intervention group) and spironolactone group (Control group).
2. Objective: To compare the antihypertensive effects and Correction of hypokalemia in patients with PA.
3. Medicine: Finerenone (10mg tablet) and the matching placebo; Spironolactone (20mg tablet) and the matching placebo.
4. Study population: Men or women aged from18 years to 75 years old, with history of hypertension, Clinic DBP <110 mmHg, SBP <180 mmHg without any antihypertensive drugs for 2 weeks, were diagnosed PA and confirmed by captopril inhibition test or Saline infusion test. At the end of induction, Serum potassium level ≥ 3 mmol/L but less than 5 mmol/L.
5. Randomized and treatment: The initial dose of finerenone group is 10mg and spironolactone group is 20mg, respectively (week 0). For patients not meeting clinic blood pressure < 140/90mmHg and the serum potassium ≥ 3.5 mmol/L, the dose of finerenone or spironolactone should be increased one tablet at every visit (week 2, week 4). The whole treatment period was 8 weeks.
6. Follow up: After the induction period of two weeks and meeting the inclusion criteria, the patients with primary aldosteronism were randomized in an equal ratio to receive finerenone 10mg once daily. Patients received the initial dose (10mg, week 0) of drug for the first two weeks of randomized treatments period. Thereafter, the dose of finernone would not be changed for the adequate blood pressure (BP) control and the normal serum potassium. For patients not meeting BP < 140/90mmHg and the serum potassium ≥ 3.5 mmol/L, the dose of finerenone would be increased to 20mg once daily for the second 2 weeks later (week 2) and 30 mg 4 weeks later (week 4), respectively. The whole treatment period was 8 weeks. if blood pressure > 160/110 mmHg during the clinical trial, amlodipine 5 mg once was added. At every visit, the clinic and ambulatory blood pressure will be measured. The levels of serum potassium, creatinine, renin, aldosterone will be examined. The urinary microalbumin creatinine ratio will be also examined.
7. Organization: The Centre for Epidemiological Studies and Clinical Trials, Department of Hypertension, Ruijin Hospital, Shanghai, China.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old.
2. History of hypertension, Clinic DBP <110 mmHg, SBP <180 mmHg without any antihypertensive drugs for 2 weeks.
3. Primary Aldosteronism diagnosed and confirmed by captopril inhibition test or Saline infusion test.
4. At the end of induction, Serum potassium level ≥ 3 mmol/L but less than 5 mmol/L.
5. Signed the informed consent

Exclusion Criteria:

1. Other kinds of secondary hypertension
2. Obesity with BMI>30kg/m²（BMI= kg/㎡）
3. Serum potassium > 5.5 mmol/L
4. Serious hypertension（msSBP≥180mmHg, and/or msDBP≥110mmHg）
5. Abnormal renal function: serum creatinine ≥ 2 × ULN or eGFR < 25 ml/(min * 1.73㎡);
6. Abnormal liver function: ALT and AST ≥ 2 × ULN；
7. Cardiac insufficiency, acute myocardial infarction, stroke or other acute cardiovascular events within 6 months;
8. Take spironolactone, guanethidine or reserpine 30 days before enrollment;
9. Known or suspected tumor; Other autoimmune diseases, uncontrolled infectious diseases, serious respiratory, blood and nervous system diseases;
10. There is a pregnancy plan in pregnancy or 3 months before and after treatment. Breast-feeding women;
11. Those who have mental illness, alcohol or drug abuse and cannot cooperate with treatment.
12. Be allergic to the study drugs
13. Without Signed the informed consent
14. Anticipating another clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-16 (Estimated); Primary Completion 2024-12-16 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
The change of 24-hour ambulatory systolic blood pressure from the baseline level. | 8 weeks
  24-hour ambulatory systolic blood pressure
The proportion of patients with normal serum potassium level. | 8 weeks
  serum potassium level

SECONDARY OUTCOMES:
The change of clinic systolic and diastolic blood pressure from the baseline level. | 8 weeks
  clinic systolic and diastolic blood pressure
The change of other components of 24-hour ambulatory blood pressure from the baseline level. | 8 weeks
  other components of 24-hour ambulatory blood pressure
The changes of plasma renin and aldosterone from the baseline levels. | 8 weeks
  plasma renin and aldosterone
The change of urinary microalbumin creatinine ratio (ACR) from the baseline level. | 8 weeks
  urinary microalbumin creatinine ratio
The change of estimate glomerular filtration rate from the baseline level. | 8 weeks
  estimate glomerular filtration rate

OTHER OUTCOMES:
Incidence of Treatment-Adverse Events as assessed by gynaecomastia, mastodynia, menstrual abnormalities, impotence, hyperkalemia and other adverse events. | 8 weeks
  gynaecomastia, mastodynia, menstrual abnormalities, impotence, hyperkalemia

CONTACTS AND LOCATIONS:
Overall Officials: Jiguang Wang, MD. PhD, Study Director — Department of Hypertension, Ruijin Hospital, Shanghai Jiaotong University School of Medicine, China
Locations (1):
- Shanghai Institite of Hypertension, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No